CLINICAL TRIAL: NCT00884143
Title: Retrospective Observational Triveneto Study on the Use of Adjuvant Hormonal Therapies in the Treatment of Hormone-responsive Breast Cancer in Two Successive Time Periods
Brief Title: Observational Triveneto Study on the Use of Adjuvant Hormonal Therapies in the Treatment of Hormone-responsive Breast Cancer
Acronym: TIME 2 CHANGE
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Raffaele Sabia MC MD, AstraZeneca
Other Study IDs: NIS-OIT-ARI-2008/1
Record Dates: First submitted 2009-04-17; First posted 2009-04-20 (Estimated); Last update posted 2010-04-20 (Estimated); Status verified 2010-04

CONDITIONS: Post Menopausal; Breast Cancer
Keywords: tamoxifen; arimidex; adjuvant hormonal therapies; breast cancer; post-menopausal; Adjuvant hormonal therapy in patients post menopausal with breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
There are different types of hormonal therapy medicines for the treatment of hormone-receptor-positive breast cancer. The purpose of this study is to determine the evolution of two types of hormonal treatment (the drug called "tamoxifen" and a group of medicines called "aromatase inhibitors") during two time periods of 12 months each, in years 2006 and 2008, in the northeast Italian regions. The study will include post-menopausal women who have initiated hormonal therapy medicines in 2006. The study will also verify the rate of implementation of the updated national and international recommendations for the use of adjuvant hormonal therapy in the hormone-receptor-positive breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal patients with surgically treated breast cancer who started adjuvant hormonal therapy between January 2006 and December 2006 or between January 2008 and December 2008
* Documented evidence of the way adjuvant hormonal treatment was initiated.

Exclusion Criteria:

* Pre- or peri-menopausal patients with surgically treated breast cancer who started adjuvant hormonal therapy
* Patients already enrolled in clinical studies aimed at investigating hormone therapies

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Post-menopausal patients with breast cancer already treated with advjuvant hormonal therapy.
Sampling Method: Non-Probability Sample
Enrollment: 515 (Actual)
Dates: Start 2009-07; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Relative frequencies of the first adjuvant hormonal treatment (tamoxifen vs aromatase inhibitor) started during two time periods of 12 months each - the years 2006 and 2008 | May-July 2009

SECONDARY OUTCOMES:
Relative frequencies of the type of initial treatment: upfront (a single drug - tamoxifen or aromatase inhibitor) or early switch (planned sequence of tamoxifen and inhibitor) | May-July 2009
Type of treatment and relative percentages of treatment undertaken by the patients after interruption of the first hormonal therapy | May - July 2009

CONTACTS AND LOCATIONS:
Overall Officials: Davide Meani, Dr., Study Chair — AstraZeneca S. p. A.; Raffaele Sabia, Study Director — AstraZeneca S.p.A
Locations (3):
- Italy (3):
  - Research Site, Aviano, PN
  - Research Site, Trento
  - Research Site, Verona